CLINICAL TRIAL: NCT00740012
Title: Blutzucker-Nachtprofile Mit Wecker Und Selbstmessungen gegenüber Fremdmessungen Durch Spezialisiertes Pflegepersonal: Eine Analyse Mittels Kontinuierlichem Glukose-Monitoring (Glucoday®)
Brief Title: Glycemic Rises After Waking Up In Response To An Alarm Clock In Type 1-Diabetic Patients Analysed With Continuous Glucose Monitoring (GlucoDay®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabeteszentrum Bad Lauterberg im Harz (Other)
Collaborators: Berlin-Chemie Menarini (Industry)
Responsible Party: Prof. Dr. Michael Nauck, Diabeteszentrum Bad Lauterberg
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Glucoday BL
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Stress; Type 1 Diabetes
Keywords: Nocturnal glucose profiles; continuous glucose profiles
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Even, low numbers (Active Comparator): They start with a alarm- clock night. No venous blood drawing.
  Interventions: Other: Continuous glucose monitoring; Other: alarm- clock intervention, patient perform blood glucose self monitoring; Other: nurse intervention; Other: Taking the patients pulse; Other: Other capillary sample
- Even, high numbers (Active Comparator): They start with a nurse performing blood glucose determination. No venous blood drawing.
  Interventions: Other: Continuous glucose monitoring; Other: alarm- clock intervention, patient perform blood glucose self monitoring; Other: nurse intervention; Other: Taking the patients pulse; Other: Other capillary sample
- Uneven, low numbers (Active Comparator): They start with an alarm- clock night and have venous blood drawing.
  Interventions: Other: Continuous glucose monitoring; Other: alarm- clock intervention, patient perform blood glucose self monitoring; Other: nurse intervention; Other: Taking the patients pulse; Other: Venous blood drawing; Other: Other capillary sample
- Uneven, high numbers (Active Comparator): They start with a nurse performing blood glucose determination and have venous blood drawing.
  Interventions: Other: Continuous glucose monitoring; Other: alarm- clock intervention, patient perform blood glucose self monitoring; Other: nurse intervention; Other: Taking the patients pulse; Other: Venous blood drawing; Other: Other capillary sample

INTERVENTIONS:
Other: Continuous glucose monitoring — Glucoday S (microdialysis system). Continuous glucose monitoring all three nights
  Other Names: Gluco Day S (Menarini Diagnostics)
Other: alarm- clock intervention, patient perform blood glucose self monitoring — Alarm clock intervention at midnight, 2 a.m., 4 a.m. and 6:45 a.m.
  Other Names: Ordinary alarm clock
Other: nurse intervention — Nurse intervention: gently drawing capillary sample (blood glucose)at midnight, 2 a.m., 4 a.m. and 6:45 a.m. .
  Other Names: professional night nurses
Other: Taking the patients pulse — In nights (a) and (b) the doctoral candidate takes the patients pulse 5-7 minutes after the alarm clock or the nurse.
  Other Names: Pulse measurment
Other: Venous blood drawing — Venous blood drawing for the determination of epinephrine, norepinephrine, cortisol, glucagon, growth hormone, and prolactin (determined by specific immunoassays at Biocientia laboratories, Jena, Germany) (6-10 minutes after midnight, 2 a.m., 4 a.m. and 6:45 a.m.)in night (a) and (b)
  Other Names: venous blood drawing from an intravenous catheter
  Arms: Uneven, high numbers; Uneven, low numbers
Other: Other capillary sample — 5-7 minutes after the alarm clock or the nurse the doctoral candidate takes another capillary sample for a laboratory glucose determination (EBIOS, Eppendorf, Hamburg, Germany) analyzer.
  Other Names: laboratory method (EBIOS, Eppendorf, Hamburg, Germany)

SUMMARY:
Study hypothesis: Waking up in response to an alarm clock may evoke a stress reaction that leads to rising glucose concentrations.

The purpose of this study was to prove this hypothesis with continuous glucose monitoring over three nights.

Night (a) with an alarm clock set at 2 h intervals for glucose self monitoring,

Night (b) with a nurse performing blood glucose determinations, and

Night (c) with the patients left undisturbed.

DETAILED DESCRIPTION:
To provide nocturnal glucose control in patients with type 1 diabetes is a therapeutic challenge. Nocturnal glucose profiles are an important tool to secure adequate glycemic control during the night. Often, patients are asked to perform self-monitoring with the help of an alarm clock. Such a recommendation depends on the accuracy of glucose concentrations determined this way. We hypothesized that alarm clocks may trigger a stressful arousal that might be accompanied by rises in glucose concentrations, consecutively leading to nocturnal glucose profiles that are not representative for undisturbed conditions.

We want to prove this hypothesis with 30 patients over three nights.

Night (a) with an alarm clock set at 2 h intervals (midnight, 2 a.m., 4a.m. and 6:45 a.m) for glucose self monitoring,

Night (b) with a nurse performing blood glucose determinations at the 2 h intervals (midnight, 2 a.m., 4a.m. and 6:45 a.m), and

Night (c) with the patients left undisturbed.

All the patients are going to use a continuous glucose monitor and half of the patients (uneven numbers) are going to have an indwelling venous cannula during night (a) and (b.

During night (a) and (b) 5-7 minutes after the scheduled times for glucose measurements the doctoral candidate is going to take the pulse, another capillary blood sample for a laboratory glucose determination (EBIOS, Eppendorf, Hamburg, Germany). Also the doctoral candidate is going to take a venous blood sample in half of the patients (uneven numbers), blood from the indwelling venous cannula for the determination of epinephrine, norepinephrine, cortisol, glucagon, growth hormone, and prolactin (determined by specific immunoassays at Biocientia laboratories, Jena, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetic patients (diagnosed longer than 2 years)
* HBA1c 5,0 - 9,5 %
* Age 18-75 years
* Hospitalized patients
* Male or female, if female exclusion of pregnancy or secure contraception
* Body-Mass-Index 19-40 kg/m²
* Patient is elucidated
* Patients agreement

Exclusion Criteria:

* Type 2-Diabetic patients or other forms of diabetes beside type 1 diabetes, diagnosed after the guidelines of the Deutsche Diabetes Gesellschaft
* HbA1c < 5,0 % or > 9,5 %
* A severe hypoglycemia with unconsciousness within the last 2 month
* Body-Mass-Index < 19 or > 40 kg/m²
* No patient agreement
* Pregnancy (positive pregnancy test) or unsecured contraception.
* Agina pectoris or acute myocardial infarct, as continuous problem
* Inadequate treated arterial hypertension > 160 mmHg systolic and/or < 95 mmHg diastolic
* Active tumor disease
* Anemia hemoglobin < 11,5 g/dl
* Treatment with steroids, sedative or anesthetics
* Infection/fewer > 37.5 °C
* Renal- malfunction (serum- creatinine > 1.5 mg/dl)
* Liver- malfunction (GPT and AP > double of upper- limit)
* Alcohol or drug abuse
* Sleep disorder
* Participation in clinical studies within the last 3 month
* Other significant health dysfunctions, which would affect the outcome of this study
* Incapable to conform the requirements of the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Glucose (continuous glucose monitoring) | 10 pm, midnight, 2 am, 4 am and 6:45 am continous glucose monitoring during three nights

SECONDARY OUTCOMES:
Hormones (norepinephrine, cortisol, glucagon, growth hormone, prolactin), Pulse, Blood glucose | 22 pm, midnight, 2 am, 4 am, 6:45 am

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, professor, Principal Investigator — Diabeteszentrum Bad Lauterberg
Locations (1):
- Diabeteszentrum Bad Lauterberg im Harz, Bad Lauterberg im Harz, Lower Saxony, Germany

REFERENCES:
- [Result] Berndt C, Köthe L, Nawrodt B, Mraz B, Patzelt-Bath A. Glycaemic rises after waking up in response to an alarm clock during the night in type 1 diabetic patients can be avoided by experienced nurses drawing blood in a hospital setting as shown by continuous glucose monitoring (GlucoDayR) (abstract 14). Diabetologia 51 (Suppl. 1): S 12
- [Derived] Berndt-Zipfel C, Kothe L, Nawrodt B, Mraz B, Patzelt-Bath A, Nauck MA. Glycaemic rises after waking up in response to an alarm clock in type 1-diabetic patients analysed with continuous glucose monitoring (GlucoDay(R) S). Exp Clin Endocrinol Diabetes. 2011 Jan;119(1):56-8. doi: 10.1055/s-0030-1265162. Epub 2011 Jan 18. PMID 21246465